CLINICAL TRIAL: NCT00028613
Title: Phase I Safety Study Of 131I-Lym-1 For The Treatment Of Previously Treated Diffuse Large B-Cell Lymphoma
Brief Title: Radiolabeled Monoclonal Antibody in Treating Patients With Previously Treated Large Cell Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRLX1400; CWRU-BRLX-1400; BRLX-303680; CWRU-090036; NCI-G01-2038
Record Dates: First submitted 2002-01-04; First posted 2003-06-30 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2014-01

CONDITIONS: Lymphoma
Keywords: recurrent adult diffuse large cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Radiation: iodine I 131 monoclonal antibody Lym-1

SUMMARY:
RATIONALE: Radiolabeled monoclonal antibodies can locate tumor cells and deliver tumor-killing substances such as radioactive iodine to them without harming normal cells.

PURPOSE: Phase I trial to study the effectiveness of radiolabeled monoclonal antibodies in treating patients who have large cell lymphoma that has been previously treated.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of iodine I 131 monoclonal antibody Lym-1 in patients with previously treated diffuse large cell lymphoma.
* Determine the safety of this drug in these patients.
* Determine the response of patients to this drug.

OUTLINE: This is a dose-escalation, multicenter study.

Patients receive unlabeled monoclonal antibody Lym-1 IV over 40 minutes followed 15-30 minutes later by iodine I 131 monoclonal antibody Lym-1 IV over 2 minutes.

Cohorts of 3-6 patients receive escalating doses of iodine I 131 monoclonal antibody Lym-1 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed weekly for 8 weeks and then every 3 months for 1 year.

PROJECTED ACCRUAL: A total of 8-36 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria

* Histologic diagnosis of B-cell diffuse large cell lymphoma (REAL classification system) confirmed by an independent central pathology reviewer.
* The tumor's B-cell phenotype will be confirmed by positive L-26 (CD20).
* Previous treatment with 2 common combination chemotherapy regimens. Patients previously treated with unlabeled monoclonal antibody therapy are eligible.
* Men or women at least 18 years of age.
* Karnofsky Performance Score (KPS) estimated to be > 60 at the time of the scheduled therapeutic dose of 131I-Lym-1.
* Life expectancy estimated to be at least 3 months from the time of the therapeutic dose of 131I Lym-1.
* Measurable disease demonstrable by physical examination or computerized tomography (CT).
* CT scan evidence of at least one indicator lesion with at least one diameter that measures > 2 cm. (The CT scan should be done within 2 weeks of the imaging study.)

Exclusion Criteria

* Inability or unwillingness to comply with the following:
* Bone marrow biopsy
* Return for follow-up visits
* Remaining motionless for extended periods of time for imaging procedures
* Serial blood/urine sampling (for dosimetry patients only)
* Pregnancy (Women of childbearing potential must be practicing an effective method of contraception.)
* Presence of a second malignancy except for basal cell skin carcinoma or carcinoma in-situ of the cervix
* Presence of active lymphomatous meningitis or other CNS involvement with lymphoma.
* HIV positive patients.
* Prior total body irradiation, or a course of prior radiation > 3,000 cGy delivered to > 20% of the central marrow or the lumbar vertebrae within 6 months of screening.
* Serum creatinine or total bilirubin > 2 x the upper limit of normal.
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT) or alkaline phosphatase > 3 x the upper limit of normal.
* Significant marrow lymphoma (defined as lymphoma cells constituting greater than 20% of the hematopoietic marrow elements from an iliac crest biopsy). A prior bone marrow biopsy is acceptable if it meets the following criteria:
* If there is prior bone marrow involvement, the biopsy must be performed within 45 days of screening.
* If there is no prior bone marrow involvement, the biopsy must be performed within 90 days of screening
* WBC count < 3,500/mm3, granulocyte count < 1,500/mm3, or platelet count < 125,000/mm3.
* Positive human anti-mouse antibodies (HAMA) serum values, defined as > 74 ng/mL at screening.
* Patients who have not recovered from toxicities of most recent anti-lymphoma therapy.
* Treatment with:
* Colony stimulating factor G-CSF or GM-CSF within 120 hours of screening laboratory assessment.
* Erythropoietin (EPO) within a month of screening laboratory assessment
* Whole blood or platelet transfusion within 120 hours of screening laboratory assessment
* History or electrocardiographic (ECG) evidence of Q-wave myocardial infarction within 6 months of screening or congestive heart failure (CHF; NYHA Stage III or IV).
* Known hypersensitivity to iodine or iodine-containing organic substances.
* Patients who require therapy with anticoagulants or antiplatelet drugs which cannot be discontinued during the study.
* Patients who are known to have antiplatelet antibodies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2001-03; Primary Completion 2001-10 (Actual); Study Completion 2001-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Omer N. Koc, MD, Study Chair — Case Comprehensive Cancer Center
Locations (1):
- Ireland Cancer Center, Cleveland, Ohio, United States